Study Title: "Manikin To Patient Intubation: Does It Translate?"

**Principal Investigator:** R. Whit Hall, M.D.

University of Arkansas for Medical Sciences 4301 W. Markham Street, Slot #512-5B

Little Rock, Arkansas 72205 Telephone: 501.603.1255

Email: HallRichardW@uams.edu

Study Location: University of Arkansas for Medical Sciences

4301 W. Markham Street Little Rock, Arkansas 72205

Date: September 19, 2017

NCT number: NCT03046966

## **Statistical Analysis**

Chi-square tests with the Benjamani-Holm p-value correction to account for test multiplicity will be used to analyze the difference in baseline measures and demographics. Chi-square testing will be utilized for comparing end of survey comfort. Logistic regression will be utilized to compare overall and first-time intubation success rates between the control and intervention groups. Logistic regression will be used to compare the difference in success rate between training level groups. To account for over-dispersion, a negative binomial regression will be utilized to assess difference in overall and first-time intubation success counts.